CLINICAL TRIAL: NCT05180734
Title: A Multicenter, Randomized, Double-Blind, Phase III Clinical Study to Evaluate the Efficacy and Safety of Toripalimab Injection Combined With Postoperative Adjuvant Chemotherapy Versus Placebo Combined With Postoperative Adjuvant Chemotherapy in Patients With Gastric or Esophagogastric Junction Adenocarcinoma After Radical Gastrectomy
Brief Title: PD1 Combined With Chemotherapy for Adjuvant Treatment of Gastric Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-045-III-GC
Record Dates: First submitted 2021-11-08; First posted 2022-01-06 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Gastric or Esophagogastric Junction Adenocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS001 240mg, Q3W with XELOX regimen or SOX regimen (Experimental): JS001 240mg, will be intravenously administered once every 3 weeks, until 17 cycles XELOX regimen (oxaliplatin + capecitabine) or SOX regimen (oxaliplatin + S-1), given in one therapeutic cycle of 3 weeks for up to 8 cycles XELOX regimen: Oxaliplatin, 130mg/m2, intravenous drip for over 3 hours, day 1, Q3W; capecitabine, 1000mg/m2, orally, twice per day, from day 1 to day 14, Q3W.
  SOX regimen: Oxaliplatin, 130mg/m2, intravenous drip for over 3 hours, day 1, Q3W; S-1 Capsules, 40-60mg, orally, twice per day, from day 1 to day 14, Q3W.
  Interventions: Biological: JS001/Placebo
- Placebo combine with chemotherapy (Placebo Comparator): XELOX regimen (oxaliplatin + capecitabine) or SOX regimen (oxaliplatin + S-1), given in one therapeutic cycle of 3 weeks for up to 8 cycles XELOX regimen: Oxaliplatin, 130mg/m2, intravenous drip for over 3 hours, day 1, Q3W; capecitabine, 1000mg/m2, orally, twice per day, from day 1 to day 14, Q3W.
  SOX regimen: Oxaliplatin, 130mg/m2, intravenous drip for over 3 hours, day 1, Q3W; S-1 Capsules, 40-60mg, orally, twice per day, from day 1 to day 14, Q3W.
  Interventions: Biological: JS001/placebo combine with Postoperative Adjuvant Chemotherapy

INTERVENTIONS:
Biological: JS001/Placebo — JS001/placebo combine with Postoperative Adjuvant Chemotherapy
  Other Names: Postoperative Adjuvant Chemotherapy
  Arms: JS001 240mg, Q3W with XELOX regimen or SOX regimen
Biological: JS001/placebo combine with Postoperative Adjuvant Chemotherapy — JS001/placebo combine with Postoperative Adjuvant Chemotherapy
  Other Names: Postoperative Adjuvant Chemotherapy
  Arms: Placebo combine with chemotherapy

SUMMARY:
This multicenter, randomized, double-blind phase III study intends to recruit about 878 patients, including PD-L1 positive 660 patients, who have received radical gastrectomy (R0 resection, D2 or more extended lymphadenectomy) with postoperative pathological stage IIB or III (AJCC Cancer Staging Manual, 8th Edition) gastric or EGJ adenocarcinoma to evaluate the efficacy and safety of JS001 combined with postoperative adjuvant chemotherapy versus placebo combined with postoperative adjuvant chemotherapy.

DETAILED DESCRIPTION:
"This is a multicenter, randomized, double-blind phase III study, plans to recruit 878 patients who received radical gastrectomy (R0, D2 or higher lymphadenectomy) with postoperative pathological stage II (T4aN0M0) or III (the 8th Edition American Joint Committee on Cancer [AJCC] Cancer Staging Manual) gastric adenocarcinoma and gastroesophageal junction adenocarcinoma, and the study intends to evaluate the efficacy and safety of JS001 combined with postoperative adjuvant chemotherapy versus placebo combined with postoperative adjuvant chemotherapy.

Patients meeting the inclusion criteria will be 1:1 randomized into JS001-chemotherapy group and placebo-chemotherapy group. The random stratification factors include adjuvant chemotherapeutic regimens (XELOX versus SOX) and tumor anatomical sites (gastric adenocarcinoma versus gastroesophageal junction adenocarcinoma).

The study treatment will be initiated 4-6 weeks after surgery, and the investigator will select XELOX (Oxaliplatin + capecitabine) or SOX (Oxaliplatin + S-1, tegafur, gimeracil and oteracil potassium) as the adjuvant chemotherapeutic regimen given as 3-week cycles for up to 8 cycles based on each patient's condition; JS001/placebo will be given for up to 17 cycles after surgery, until intolerable toxicity, disease recurrence, patient's withdrawal of consent, investigator's judgment that the patient needs to be withdrawn from the study treatment, or death, whichever comes first.

Safety evaluation, including vital signs, ECOG score, physical examination and laboratory examinations, will be performed on a regular basis during the treatment.

This study will end after the main analysis node of DFS and unblinding for analysis are achieved, or 5 years after enrollment of the last patient, whichever comes first. The Sponsor is entitled to terminate the study at any time due to specific reasons (e. g, major safety issues, force majeure, etc.).

Radiological follow-up: tumor response evaluation will be performed once every 12 weeks ±7 days within the first 5 years after randomization, and once per year subsequently, until disease recurrence or death. When symptoms or signs of suspected recurrence/metastasis occur, the radiological evaluation can be performed at any time. Disease recurrence is defined as local recurrence or distant metastases with clear radiological evidence (CT or MRI).

Survival follow-up: it will be performed once every 12 weeks after disease recurrence, until patient's withdrawal of informed consent, loss to follow-up or death, whichever comes first.

Safety follow-up: adverse events will be closely followed up and recorded, until 60 days after the last dose of treatment or the end of study follow-up (death, loss to follow-up, withdrawal of consent form and the end of study), whichever comes first.

"

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 18-75 years.
2. No residual tumor (R0) after D2 or greater lymphadenectomy through laparotomy.
3. According to the definition of the 8th edition of the AJCC Cancer Staging Manual, patients with gastric adenocarcinoma confirmed by histopathology, pathological stage II (T4aN0M0) and stage III, including gastroesophageal junction adenocarcinoma (GEJ) patients.
4. Patients need to provide sufficient formalin-fixed paraffin-embedded (FFPE) neoplasm tissue specimens or sections that are confirmed to be PD-L1 positive (CPS ≥ 1) by lab test at the central laboratory.
5. ECOG performance status 0-1.
6. No metastasis or recurrence as radiologically confirmed.
7. Patients must have adequate organ function as assessed in the laboratory tests.
8. Patients must provide informed consent for this study, and sign the written informed consent form voluntarily before the initiation of the study, and are willing and able to comply with the scheduled visits, treatment plan, laboratory examinations and other study procedures in the study.
9. Female patients of childbearing age must take a serum pregnancy test within 7 days before randomization with negative results, and agree to adopt reliable and effective contraceptive methods during the study.

EXCLUSION CRITERIA

1. Previous use of non-surgical therapy (e.g., radiotherapy, chemotherapy, hormone therapy) for gastric adenocarcinoma.
2. Having liver, peritoneal or other distant metastasis.
3. Having malignant tumors other than gastric adenocarcinoma within 5 years before randomization.
4. Pevious treatment targeting PD-1 receptor or its ligand PD-L1 or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) receptor;
5. Previous history of serious allergy to monoclonal antibody or other biological preparations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
DFS in the PD-L1-positive population evaluated by the BICR | 5 years
  To evaluate the disease-free survival (DFS) by the blind independent central review (BICR) for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in PD-L1-positive patients with gastric or GEJ adenocarcinoma after radical gastrectomy.

SECONDARY OUTCOMES:
OS in the PD-L1-positive population | 5 years
  To evaluate the OS for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in PD-L1-positive patients with gastric or gastroesophageal junction adenocarcinoma after radical gastrectomy.Toripalimab Injection (JS001) combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in patients with gastric or gastroesophageal junction adenocarcinoma after radical gastrectomy.
DFS in the PD-L1-positive population evaluated by the investigator | 5 years
  To evaluate the disease-free survival (DFS) by the investigator for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in PD-L1-positive patients with gastric or GEJ adenocarcinoma after radical gastrectomy.
DFS in the ITT population evaluated by the BICR and investigator, respectively | 5 years
  To evaluate the disease-free survival (DFS) by the blind independent central review (BICR) and investigator,respectively, for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in the ITT population.
OS in the ITT population | 5 years
  To evaluate the OS for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in the ITT population.
DFS rate at 3 years in the PD-L1-positive population and the ITT population evaluated by the BICR and investigator, respectively | 3 years
  To evaluate the disease-free survival (DFS) rate at 3 years by the BICR and investigator, respevtively, for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in the PD-L1-positive population and the ITT population.
DFS rate at 5 years in the PD-L1-positive population and the ITT population evaluated by the BICR and investigator, respectively | 5 years
  To evaluate the disease-free survival (DFS) rate at 5 years by the BICR and investigator, respevtively, for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in the PD-L1-positive population and the ITT population.
OS rate at 3 years in the PD-L1-positive population and the ITT population | 3 years
  To evaluate the OS rate at 3 years for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in the PD-L1-positive population and the ITT population.
OS rate at 5 years in the PD-L1-positive population and the ITT population | 5 years
  To evaluate the OS rate at 5 years for toripalimab combined with adjuvant chemotherapy versus placebo combined with adjuvant chemotherapy in the PD-L1-positive population and the ITT population.
Immunogenicity of toripalimab | Up to the 90 days from last dose of toripalimab
  To evaluate the incidence and titer of anti-drug antibody (ADA) of toripalimab, and further analyze ADA-positive samples for the presence of Neutralising antibodies (Nab).
Blood trough concentration of toripalimab | Up to the 90 days from last dose of toripalimab
  To evaluate the blood trough concentration of toripalimab

CONTACTS AND LOCATIONS:
Locations (71):
- China (71):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Peple's Hospital of Chizhou, Chizhou, Anhui
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking University People's hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - The first affiliated hospital of chongqing medical universit, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - The first Hospital of Lanzhou University, Lanzhou, Gansu
  - Wuwei Cancer Hospital of Gansu Province, Wuwei, Gansu
  - Guandong General Hospital, Guangzhou, Guandong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guandong
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The First Affiliated Hospital of Sun yat-sen University, Guangzhou, Guangdong
  - Affiliated Cancer Hospital and Institute of Ghuangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The 2ed Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - Henan cancer hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hopital, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu cancer hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second People's Hospital of Wuxi, Wuxi, Jiangsu
  - Jiangmen Central Hospital, Nanchang, Jiangxi
  - The first Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shengyang, Liaoning
  - LiaoNing Cancer Hospital & Institute, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai University Affiliated Hosptial, Xining, Qinghai
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao central medical group, Qingdao, Shandong
  - Jinan Central Hospital, Jinan, Shangdong
  - Shandong Provincial Hospital, Jinan, Shangdong
  - Affiliated Hospital of Jining Medical University, Jining, Shangdong
  - Zhongshan Hospital, Fudan university, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Tangdu hospital, Air force Military Medical University, Xian, Shanxi
  - Xijing hospital, Air force Military Medical University, Xian, Shanxi
  - SiChuan Cancer Hospital, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Cancer Hospital affiliated to Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The first affiliated hospital of Zhejiang medical university, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang